CLINICAL TRIAL: NCT05223686
Title: A Phase I Clinical Study To Evaluate the Safety and Tolerability of Human CD19-CD22 Targeted T Cells Injection for In Subjects With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia.
Brief Title: To Evaluate the Safety and Tolerability of Human CD19-CD22 Targeted T Cells Injection for Subjects With R/R B-ALL.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-ALL02
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; CD19-CD22; CAR-T; relapsed/refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human CD19-CD22 Targeted T Cells Injection (Experimental): Single administration：1.0×10^6 CAR+T, 3.0×10^6 CAR+T，6.0×10^6 CAR+T
  Interventions: Drug: Human CD19-CD22 Targeted T Cells Injection

INTERVENTIONS:
Drug: Human CD19-CD22 Targeted T Cells Injection — One time single predetermined dose level CAR-positive T cells will be utilized based on the NMPA approved product label.
  Other Names: CD19-CD22 CAR-T

SUMMARY:
To evaluate the safety and tolerability of Human CD19-CD22 Targeted T Cells Injection for the treatment of Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia. Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of CD19-CD22 CAR+ T cells.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation phase I clinical study to explore the safety, tolerability and pharmacokinetic characteristics of Human CD19-CD22 Targeted T Cells Injection. To preliminary observe the effect of Human CD19-CD22 Targeted T Cells Injection in relapsed/refractory B-cell acute lymphoblastic leukemia, and to explore the clinically applicable dose and reinfusion regimen for phase II.

Participants with relapsed/refractory B-cell Acute Lymphoblastic Leukemia can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, Electrocardiograph, Computedtomography （CT）/ Magnetic Resonance Imaging(MRI) / Positron Emission Tomography（PET）, and blood draws. Participants receive chemotherapy prior to the infusion of CD19-CD22 CAR+ T cells. After the infusion, participants will be followed for side effects and effect of CD19-CD22 CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia:

* 18~70 years old (including cut-off value), male and female;
* Expected survival > 12 weeks;
* ECOG score 0-1;
* Bone marrow examination clearly diagnosed as B-cell acute lymphoblastic leukemia , CD19 or/and CD22 positive , and who met one of the following conditions:

  1. Those who failed to achieve CR after at least 2 courses of standard chemotherapy or had early relapse after complete remission (<12 months) or late relapse after complete remission (≥ 12 months) and failed to achieve CR after 1 course of standard chemotherapy;
  2. For Ph+ ALL: in addition to receiving at least 2 courses of standard chemotherapy, at least two TKIs should be treated with no complete remission or relapse after complete remission; (Patients who cannot tolerate TKI therapy or have TKI treatment contraindications or have T315i mutation are excluded);
  3. Those who relapse after stem cell transplantation are not affected by previous treatments;
* The venous access required for collection can be established and mononuclear cell collection can be determined by the investigators;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Serum creatinine≤1.5×ULN;
  2. Left ventricular ejection fraction>50%;
  3. Baseline blood oxygen saturation>96%;
  4. Total bilirubin≤2×ULN; ALT and AST≤3×ULN (As judged by the investigator, the elevation of transaminase caused by the ALL disease itself, ALT and AST≤5×ULN);
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

Any one of the following conditions cannot be selected as a subject：

* Graft-versus-host disease (GVHD), or need to use immunosuppressants after transplantation;
* Patients with hyperleukocytosis (white blood cell count ≥50×10^9/L) or whose disease progressed rapidly according to the investigator's judgment at the time of enrollment and cannot ensure the completion of a complete treatment cycle;
* Malignant tumors other than acute lymphoblastic leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection and thyroid cancer after radical resection ;
* Subjects with positive HBsAg or HBcAb and peripheral blood HBV DNA titer detection higher than the lower limit of the research center can detect; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; syphilis positive;
* Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
* Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* Received CAR-T treatment or other gene therapies before enrollment;
* Patients with symptoms of central nervous system;
* Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use);
* The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) | 28 days post infusion
  Safety indicators

SECONDARY OUTCOMES:
Adverse events； | 28 days post infusion
  Safety indicators
Pharmacokinetic parameters: the highest concentration of anti-human CD19-CD22 T cells amplified in peripheral blood after reinfusion; | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Pharmacokinetic parameters: the time to reach the highest concentration of anti-human CD19-CD22 T cells amplified in peripheral blood after reinfusion; | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Pharmacokinetic parameters: the 28-day area under the curve of anti-human CD19-CD22 T cells amplified in peripheral blood after reinfusion; | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Pharmacodynamic parameters: the detection counts of CD19 or CD22 positive B cells in peripheral blood; | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Pharmacodynamicparameters: the detection values of IL-6, CRP, and IL-15 cytokines in peripheral blood; | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Overall response rate (ORR) after administration | 3 months post infusion
  Effectiveness Metrics
Duration of remission (DOR) after administration | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Progress Free Survival (PFS) after administration | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
Overall Survival (OS) after administration | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Effectiveness Metrics
The immunogenicity of Human CD19-CD22 Targeted T Cells Injection. (the detection of human anti-mouse antibody) | 2 years post infusion（the last subject will be followed up to 15 years after infusion）
  Safety indicators

CONTACTS AND LOCATIONS:
Overall Officials: Jianqing Mi, Doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No